CLINICAL TRIAL: NCT02780401
Title: A Phase I Trial of the Safety and Immunogenicity of a DNA Plasmid Based Vaccine (WOKVAC) Encoding Epitopes Derived From Three Breast Cancer Antigens (IGFBP-2, HER2, and IGF-1R) in Patients With Breast Cancer
Brief Title: Vaccine Therapy in Preventing Cancer Recurrence in Patients With Non-Metastatic, Node Positive, HER2 Negative Breast Cancer That is in Remission
Acronym: WOKVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Professor, Clinical Research Division, National Cancer Institute (NCI)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9626; NCI-2016-00581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UW14090; N01-CN-2012-00033; UWI4090 (Other: University of Wisconsin Hospital and Clinics); UWI2014-03-01 (Other: DCP); N01CN00033 (NIH); P30CA014520 (NIH); RG1716053 (Other: Fred Hutch/University of Washington Cancer Consortium); NCT03156309 (obsolete NCT alias)
Record Dates: First submitted 2016-04-27; First posted 2016-05-23 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: HER2/Neu Negative; No Evidence of Disease; One or More Positive Axillary Nodes; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: Stage I; Stage II; Stage III
MeSH Terms: conditions — Breast Neoplasms | interventions — sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (WOKVAC with sargramostim) (Experimental): Patients receive WOKVAC with sargramostim ID on day 1. Courses repeat every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients with ALND will have vaccine administered to the contralateral arm. Patients with bilateral ALND will have vaccine administered in the thigh. As much as possible each vaccine dose will be given within the same draining lymph node site. Patients will be monitored for a minimum of 60 minutes post vaccine administration.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: pUMVC3-IGFBP2-HER2-IGF1R Plasmid DNA Vaccine; Biological: Sargramostim

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: pUMVC3-IGFBP2-HER2-IGF1R Plasmid DNA Vaccine — Given ID
  Other Names: pUMVC3-IGFBP2-HER2-IGF1R; pUMVC3-IGFBP2-HER2-IGF1R Vaccine; WOKVAC; WOKVAC Vaccine
Biological: Sargramostim — Given ID
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase I trial studies the side effects and best dose of a vaccine therapy in preventing cancer from coming back in patients with non-metastatic, node positive, human epidermal growth factor receptor (HER)2 negative breast cancer in which all signs and symptoms have disappeared. Vaccines made from deoxyribonucleic acid (DNA) may help the body build an effective immune response to kill tumor cells. Giving multiple vaccinations may make a stronger immune response and prevent or delay the return of cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a dose escalation study of WOKVAC.

Patients receive WOKVAC with sargramostim intradermally (ID) on day 1. Courses repeat every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients with axillary lymph node dissection (ALND) will have vaccine administered to the contralateral arm. Patients with bilateral ALND will have vaccine administered in the thigh. As much as possible each vaccine dose will be given within the same draining lymph node site. Patients will be monitored for a minimum of 60 minutes post vaccine administration.

After completion of study treatment, patients are followed up at 1 month, 6 months and annually for up to 5 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-metastatic, node positive, HER2 negative breast cancer, confirmed by pathology report, who are in remission and defined as having no evidence of disease (NED); HER2 negative is defined as

  * 0-1+ HER2 expression by immunohistochemistry (IHC) OR
  * Fluorescence in situ hybridization (FISH) negative OR
  * HER2 2+ and FISH negative
* Patients must be at least 28 days post cytotoxic chemotherapy, radiotherapy, monoclonal antibody and/or other biologic therapy, prior to enrollment; patients on bisphosphonates, denosumab, and/or endocrine therapy administered during the study are eligible and may continue throughout duration of study
* Patients must be at least 28 days post systemic steroids prior to enrollment
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status score of =< 2
* White blood cell (WBC) >= 3000/mm^3
* Hemoglobin (Hgb) >= 10 g/dl
* Lymphocyte count >= 800/mm^3
* Platelet count >= 75,000/mm^3
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min
* Total bilirubin =< 1.5 mg/dl
* Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT) =< 2 times upper limit of normal (ULN)
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* The effects of WOKVAC on the developing human fetus are unknown. For this reason, patients who are having sex that can lead to pregnancy must agree to use adequate contraception (hormonal, barrier method of birth control, or abstinence) for the duration of study participation; should a woman become pregnant while participating in the study, she should inform her study doctor immediately and will not receive any more study treatment
* Left ventricular ejection fraction (LVEF) results must be >= lower limit of normal (LLN) for institution performing based on results from the multi-gated acquisition (MUGA) or echocardiogram (ECHO) done at baseline
* Willing to not undergo any elective surgical procedure with general anesthesia or conscious sedation through the 1 month post-vaccination visit
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Dilated cardiomyopathy
  * Unstable angina within 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
  * Symptomatic pericardial effusion
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to WOKVAC
* Patients with any contraindication or known hypersensitivity to receiving sargramostim (recombinant human granulocyte macrophage colony stimulating factor [rhuGM-CSF]) or other yeast based products
* Pregnant women are excluded from this study because WOKVAC is a vaccine agent with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with WOKVAC breastfeeding should be discontinued if the mother is treated with this vaccine
* History of diabetes
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* History of autoimmunity that has not been controlled with treatment in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2022-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
The original intent of this study did not define a plan to make IPD available. We will follow the NCI policy.

REFERENCES:
- [Result] Disis ML, Gad E, Herendeen DR, Lai VP, Park KH, Cecil DL, O'Meara MM, Treuting PM, Lubet RA. A multiantigen vaccine targeting neu, IGFBP-2, and IGF-IR prevents tumor progression in mice with preinvasive breast disease. Cancer Prev Res (Phila). 2013 Dec;6(12):1273-82. doi: 10.1158/1940-6207.CAPR-13-0182. Epub 2013 Oct 23. PMID 24154719

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim; Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim; Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim: Patients receive WOKVAC with sargramostim ID on day 1. Courses repeat every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients with ALND will have vaccine administered to the contralateral arm. Patients with bilateral ALND will have vaccine administered in the thigh. As much as possible each vaccine dose will be given within the same draining lymph node site. Patients will be monitored for a minimum of 60 minutes post vaccine administration.
Period: Overall Study
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
Started | 10 | 12 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: This study allowed for replacement of patients that did not complete the 3 WOKVAC vaccines + the 1 month post vaccine 3 visit.
Groups:
- Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim; Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim; Reatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim: Patients receive WOKVAC with sargramostim ID on day 1. Courses repeat every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients with ALND will have vaccine administered to the contralateral arm. Patients with bilateral ALND will have vaccine administered in the thigh. As much as possible each vaccine dose will be given within the same draining lymph node site. Patients will be monitored for a minimum of 60 minutes post vaccine administration.
  Laboratory Biomarker Analysis: Correlative studies
  pUMVC3-IGFBP2-HER2-IGF1R Plasmid DNA Vaccine: Given ID
  Sargramostim: Given ID
- Total: Total of all reporting groups
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Reatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim | Total
Number analyzed (Participants) | 10 | 12 | 10 | 32
Age, Continuous [Mean (Full Range); unit: years] | 51 [37 to 64] | 53 [31 to 64] | 45 [36 to 79] | 51.9 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 9 | 31
  Male | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Non Hispanic Latino | 10 | 10 | 8 | 28
  White - Hispanic or Latino | 0 | 1 | 0 | 1
  White - Not Reported | 0 | 1 | 0 | 1
  Asian - Unknown | 0 | 0 | 1 | 1
  Unknown - Unknown | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 10 | 30
  Canada | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Per Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicities by grade that were related (possibly, probably or definitely) to the study vaccine noted during the immunization regimen will be summarized. This is done by arm, Grade and Attribution to study vaccine.
Time Frame: Up to 9 months
Measure: Number; unit: Count of Related Adverse Events per Arm
Units Other Than Participants: Count of Related Adverse Events per Arm
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
Number analyzed (Participants) | 10 | 12 | 10
Number analyzed (Count of Related Adverse Events per Arm) | 47 | 54 | 37
Count of Related Adverse Events per Arm
  Grade 1 related adverse events | 45 | 53 | 30
  Grade 2 related adverse events | 2 | 1 | 7

2. Secondary Outcome: Assessment of IgG Antibodies
Description: Immune response will be measured by indirect enzyme-linked immunosorbent assay and serum antibody avidity to determine an avidity index before and after vaccination. Patients will be considered to have developed an antibody response if antigen specific IgG antibodies are both detectable and have moderate to high avidity.
Time Frame: Up to 4 months
Reporting Status: Not Posted

3. Secondary Outcome: Assessment of T Helper Th1:Th2 Ratio
Description: IFN-g (Th1) and IL-10 (Th2) T-cells will be evaluated using enzyme-linked immunosorbent spot assay. Patients will be considered to have developed a Th1 immune response as the sum IFN-Ɣ magnitude from all antigens to maximum response. This will be presented as a median fold change from baseline to the maximum response (1 or 6 months after vaccination).
Time Frame: Up to 9 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
Number analyzed (Participants) | 10 | 9 | 10
score on a scale | 3.5 [1.3 to 667] | 4.5 [-1.3 to 1377] | 1.2 [-3.8 to 5.7]

4. Secondary Outcome: Assessment of the Immunogenicity of WOKVAC by Generation of IGFBP-2, HER2, and IGF-1R Specific Type 1 (Th1) T- Cells
Description: Immune responses will be measured by IFN-g enzyme-linked immunosorbent spot assay using blood (PBMC) represented by a maximum immune response generated to each antigen individually measured as corrected spots per well (cSPW). At the immune evaluations, each patient was given a value to indicate their immune response at both baseline and post vaccination. This data is represented by a median response, at both baseline (before vaccination) and 1 month or 6 months after the last vaccination of 3 vaccines (maximum response), to each of the 3 vaccine antigens HER2, IGFBP-2 or IGF1R.
Time Frame: Up to 24 weeks
Measure: Median (Full Range); unit: correct spots per well (cSPW)/10^6 PBMC
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
Number analyzed (Participants) | 10 | 10 | 10
correct spots per well (cSPW)/10^6 PBMC
  HER2 - Baseline | 92 [2.5 to 1276] | 109 [0 to 1218] | 402 [92 to 1540]
  HER2 - Maximum | 639 [14 to 1695] | 203 [10 to 1034] | 237.5 [0 to 1517]
  IGF-1R - Baseline | 0 [0 to 0] | 0 [0 to 508] | 107 [0 to 477]
  IGF-1R - Maximum | 0 [0 to 116] | 18 [0 to 507] | 76 [5.6 to 1172]
  IGFBP-2 - Baseline | 58.5 [0 to 868] | 179 [0 to 490] | 123 [0 to 890]
  IGFBP-2 - Maximum | 184.5 [2.8 to 661] | 215 [16 to 459] | 207.5 [7.5 to 355]

5. Secondary Outcome: Level of Antigen Specific Central and Effector Memory Phenotypes (Persistent Memory T Cell Response)
Description: Assessed by flow cytometry of peripheral blood mononuclear cells using an established T-cell activation panel and summarized with mean and standard deviation or median and range over time.
Time Frame: Up to 6 months after the last vaccine
Reporting Status: Not Posted

6. Secondary Outcome: Modulation of Myeloid Derived Suppressor Cell Levels
Description: Assessed by flow cytometry of peripheral blood mononuclear cells using an established myeloid derived suppressor cell/ regulatory T-cell panel and summarized with mean and standard deviation or median and range over time.
Time Frame: Up to 24 weeks
Measure: Median (Full Range); unit: percentage of m-MDSC
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
Number analyzed (Participants) | 9 | 10 | 9
percentage of m-MDSC | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.08] | 0.01 [0.00 to 0.09]

7. Secondary Outcome: Modulation of T Regulatory Cell Levels
Description: Assessed by flow cytometry of peripheral blood mononuclear cells using an established myeloid derived suppressor cell/ regulatory T-cell panel and summarized with median and range. FOXP3 is used to identify regulatory T cells, specifically CD4+ cells isolated from PBMC.
Time Frame: Up to 24 weeks
Measure: Median (Full Range); unit: % of Foxp3+ cells among CD4+ cells
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
Number analyzed (Participants) | 9 | 10 | 9
% of Foxp3+ cells among CD4+ cells | 8 [3 to 9] | 5 [3 to 8] | 4 [3 to 7]

ADVERSE EVENTS:
Time Frame: Adverse events including Serious Adverse Events (SAEs) will be collected through the 6 month follow-up visit (total of 9 months). This is the incidence of all reported adverse events regardless of attribution.
Arm/Group | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/12 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 12/12 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (WOKVAC With Sargramostim) - Dose 150 mcg + 100 mcg Sargramostim (N=10) | Treatment (WOKVAC With Sargramostim) - Dose 300 mcg + 100 mcg Sargramostim (N=12) | Treatment (WOKVAC With Sargramostim) - Dose 600 mcg + 100 mcg Sargramostim (N=10)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) — Arm 1 - 1/2 was deemed possibly related to study treatment Arm 3 - 1/1 was deemed probably related to study treatment
Alanine aminotransferase increased (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) — Arm 1 - 1/1 was deemed possibly related to study treatment Arm 2 - 2/2 deemed possibly related to study treatment
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Alanine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) — Arm 3 - 1/2 was possibly related to the study treatment as it increased in grade (in the same patient)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Allergic reaction was unrelated to the study vaccine
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) — Arm 1 - 1/2 events was deemed possibly related as it changed in grade
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Chest pain was unrelated to study vaccine
Chills (General disorders) | 4 (5) | 5 (8) | 0 (0) — Arm 1 - 3/5 events were deemed related to the study treatment Arm 2 - 5/8 events were deemed related to the study treatment
Constipation (Gastrointestinal disorders) | 3 (5) | 2 (2) | 1 (1) — Arm 1 - 3/5 events were deemed possibly related to study treatment
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 5 (7) — Arm 2 - 1/5 events was deemed possibly related to study treatment
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) — Arm 3 - 1/3 events was deemed possibly related to treatment
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) — Arm 2 - 1/1 events was deemed possibly related to study treatment Arm 3 - 1/2 events was deemed possibly related to study treatment
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) — Arm 2 - 1/3 events was deemed probably related to study treatment Arm 3 - 1/2 events was deemed possibly related to study treatment
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Erythema multiforme is unrelated to the study vaccine
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Arm 3 - 1/1 events was deemed possibly related to study treatment
Eye Disorder - Other (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Eye disorder was unrelated to study vaccine
Fatigue (General disorders) | 5 (8) | 3 (4) | 1 (1) — Arm 1 - 6/8 events were deemed related to study treatment Arm 2 - 4/4 events were deemed related to study treatment Arm 3 - 1/1 events was deemed possibly related to study treatment
Flu like symptoms (General disorders) | 5 (6) | 8 (11) | 2 (2) — Arm 1 - 6/6 events were deemed related to study treatment Arm 2 - 10/11 events were deemed related to study treatment Arm 3 - 2/2 events were deemed related to study treatment
Flushing (Vascular disorders) | 2 (4) | 2 (2) | 0 (0) — Arm 1 - 4/4 events were deemed possibly related to study treatment Arm 2 - 1/2 events was deemed possibly related to study treatment
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 4 (10) | 3 (3) — Arm 1 - 1/5 events was deemed possibly related to study treatment Arm 2 - 4/10 events was deemed possibly related to study treatment Arm 3 - 1/3 events was deemed possibly related to study treatment
Hot flashes (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Glucose (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 2 (2) — Arm 2: 2/4 glucose results were deemed possibly related to the study vaccine
Hypertension (Vascular disorders) | 7 (11) | 2 (2) | 1 (1) — Note: Hypertension was defined as a reported abnormal blood pressure per protocol
Hyperthyroidism (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) — Arm 3 - 1/1 events was deemed possibly related to study treatment
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 3 (3) — Arm 1 - 1/5 events was deemed possibly related to the study treatment Arm 2 - 1/2 events was deemed possibly related to the study treatment Arm 3 - 1/3 events was deemed possibly related to the study treatment
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) — Arm 1 - 1/1 events is deemed possibly related to study treatment
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (3) — Arm 2 - 2/3 events was deemed possibly related to study treatment Arm 3 - 1/3 events was deemed possibly related to study treatment
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) — Arm 1 - 1/1 adverse event was deemed possibly related to study vaccination
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 9 (14) | 10 (17) | 7 (13) — Arm 1 - 12/14 events were deemed related to the study treatment Arm 2 - 14/17 events were deemed related to the study treatment Arm 3 - 12/13 events were deemed related to the study treatment
Investigations - Other (Investigations) | 1 (1) | 0 (0) | 0 (0)
Complement 3 (Investigations) | 0 (0) | 2 (2) | 2 (2) — Arm 2 - 1/2 events was deemed possibly related to study treatment
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Arm 1 - 1/1 events was deemed probably related to the study treatment
Lymphocyte count decreased (Investigations) | 7 (7) | 4 (4) | 5 (5) — Arm 1 - 2/7 events was deemed possibly related to study treatment Arm 2 - 2/4 events was deemed possibly related to study treatment Arm 3 - 2/5 events was deemed possibly related to study treatment
GAD65 (Investigations) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
ANA (Investigations) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0) — Arm 2 - 2/2 events were deemed probably related to study treatment
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 6 (7) | 1 (1) — Arm 1 - 3/7 events was deemed possibly related to study treatment Arm 2 - 3/7 events was deemed possibly related to study treatment
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (11) | 3 (3) | 3 (3) — Arm 1 - 4/11 events was deemed possibly related to study treatment Arm 2 - 1/3 events was deemed possibly related to study treatment Arm 3 - 1/3 events was deemed possibly related to study treatment
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) — Arm 1 - 1/1 events was deemed possibly related to study treatment Arm 2 - 1/1 events was deemed possibly related to study treatment Arm 3 - 1/1 events was deemed possibly related to study treatment
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (5) | 1 (1) | 1 (3) — Arm 1 - 1/5 events was deemed possibly related to study treatment Arm 2 - 1/1 events was deemed possibly related to study treatment Arm 3 - 1/3 events was deemed possibly related to study treatment
Pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Arm 1 - 1/1 events was deemed possibly related to study
Phantom pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) — ARM 2: 1/2 palpitations was deemed possibly related to study vaccine and was a Grade 1
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) — Arm 3 - 1/2 events was deemed possibly related to study treatment
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (6) | 2 (2) — Arm 1 - 1/5 events was deemed possibly related to study treatment Arm 2 - 1/6 events was deemed possibly related to study treatment Arm 3 - 1/2 events was deemed possibly related to study treatment
Presyncope (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) — Arm 3 - 2/2 events was deemed possibly related to study treatment
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (2) — Arm 2 - 2/3 events was deemed possibly related to study treatment Arm 3 - 1/2 events was deemed possibly related to study treatment
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 2 (3) | 0 (0) | 1 (1) — ARM 1: 1 patient: replacement of breast implants 1 patient: revision of DIEP flap reconstruction and delayed recovery from anesthesia
Upper respiratory infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Urinary tract infection (UTI) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) — Arm 1 - 1/2 events was deemed possibly related to study treatment
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 5 (5) | 6 (7) | 4 (4) — Arm 1 - 1/5 events was deemed possibly related to study treatment Arm 2 - 2/7 events was deemed possibly related to study treatment Arm 3 - 3/4 events was deemed possibly related to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02780401/Prot_SAP_000.pdf